CLINICAL TRIAL: NCT05744492
Title: Effects of a Multicomponent Exercise Program on the Intrinsic Capacity of Community-dwelling Older Adults Under the ICOPE Framework: Study Protocol for a Multi-center Randomized Control Trial in Primary Care
Brief Title: Multicomponent Exercise Program on the Intrinsic Capacity (ICOPE) of Community-dwelling Older Adults in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: European University Spain (Other)
Collaborators: Public Health Service of Madrid (Other)
Responsible Party: Principal Investigator, Maria-Jose Gimenez Mestre, Principal Investigator, Physical Therapy & Health Sciences Research Group, Adjunct lecturer, European University Spain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22/574
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Healthy Ageing
Keywords: Frail Older Adults; Elderly; Primary care; Physical Therapy

STUDY DESIGN:
Intervention Model Description: Three-branch multi-center randomized clinical trial with 1:1:1 allocation to a center-based supervised Vivifrail MCE, a home-based non-supervised Vivifrail MCE program, or to a control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Physical therapists in charge of the intervention will not be endpoint's evaluators. Participants will be informed and encouraged not to disclose their assignment to the endpoints' evaluators, which will remain blinded to individual's membership. Investigators responsible for the statistical analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Vivifrail (S-ViF) (Experimental): A 12-week intervention program that consists of walking every day (the time is individually adjusted) and exercising 3 times a week. Shared features of the different programs are the inclusion of resistance, cardiovascular, balance and flexibility components. All exercises will be individually tailored. Once-per-week, subjects assigned to this group will attend the primary care center to execute one of the three exercise sessions per week under the supervision of the physical therapist.
  Interventions: Other: Vivifrail multicomponent exercise program
- Non-supervised Vivifrail Group (NS-ViF) (Experimental): A 12-week intervention program that consists of walking every day (the time is individually adjusted) and exercising 3 times a week. Shared features of the different programs are the inclusion of resistance, cardiovascular, balance and flexibility components. All exercises will be individually tailored. Subjects assigned to this group will follow a domiciliary-based program and they will not attend the primary care center to execute the exercises.
  Interventions: Other: Vivifrail multicomponent exercise program
- Control group (UCG) (No Intervention): Subjects will receive usual care following prevention protocols of Primary Care Services in Madrid. Concisely, the benefits of physical activity are individually explained and subjects are advised to walk as much as possible with the aim of reaching at least 30 minutes a day, 5 days a week, following the recommendations of the World Health Organization. No structured exercise-based interventions are programmed in this group.

INTERVENTIONS:
Other: Vivifrail multicomponent exercise program — Resistance: 3 sets of 2 repetitions of 3-4 exercises with a 1 to 3-minute break between sets. Intensity from 30-repetition maximum (RM) at weeks 1-6 to 20-RM at weeks 7-12.
  Balance training: both static and dynamic. Subjects will increase the number of repetitions, the difficulty of the exercises or will add external perturbations to the tasks (unstable surfaces, obstacles, or visual deprivation) along the duration of the interventions to guaranteeing progression. In the case of high risk of falling the number, frequency and volume of balance exercises will be increased.
  Flexibility: a set of stretching exercises at the end of each session. Subjects will be instructed to stretch until they feel tension in their muscles without reaching discomfort. Stretching will be maintained for 10 sec. and repeated 2-3 times.
  Cardiovascular: walking-based activities oriented to increase cardiorespiratory fitness. They will range from 5-10 sec. to 45 min/session.
  Arms: Non-supervised Vivifrail Group (NS-ViF); Supervised Vivifrail (S-ViF)

SUMMARY:
A three-branch multi-center randomized clinical trial to be conducted in 6 public Primary Care centers located in the city of Madrid (Spain). A total of 180 older adults (>=70 years old) presenting with declines in the intrinsic capacity (IC) locomotion domain will be recruited in the participating centers. They will be randomized in a 1:1:1 ratio to a center-based supervised Vivifrail multicomponent exercise (MCE) program, a home-based non-supervised Vivifrail MCE program, or to a control group. The intervention consists of thrice-a-week exercise sessions encompassing strength, aerobic, flexibility, and balance and gait training tailored to the individual's baseline functional ability. IC will be assessed through its operational domains following ICOPE guidelines at baseline and 6 and 12 weeks after the start of the intervention. Secondarily, effects on frailty status and health-related quality of life will be evaluated.

This study might bring new evidence around the ICOPE recommendation on the Vivifrail MCE for the management of IC locomotion declines in Primary Care for the first time. Gaining insight on exercise interventions for IC promotion/maintenance will reinforce current recommendations and contribute to the development of real-world strategies for healthy aging promotion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years old
* Attending participating primary care centers
* Pre-frailty or frailty according to Fried's criteria
* SPPB <10
* Barthel Index Score ≥60
* Being able to communicate and ambulate with or without technical aids
* Relative/caregiver willingness to supervise the exercise (if needed)

Exclusion Criteria:

* Major cognitive disorder according to the Diagnostic and Statistical Manual of Mental Disorders V criteria or the Global Deterioration Scale by Reisberg (GDS>4)
* Physically active individuals (moderate-to-vigorous physical activity greater than 150 minutes per week according current physical activity guidelines for older adults) or those already participating in structured physical exercise programs
* Diagnosis of a terminal illness/life expectancy ≤3months
* Lack of possibility of follow-up
* Institutionalized or awaiting institutionalization
* Any contraindications for physical exercise or testing procedures, including but not limited to: myocardial infarction in the past 6 months; unstable angina pectoris; uncontrolled arrhythmia; unstable cardiovascular disease or other unstable medical condition; uncontrolled arterial hypertension; recent pulmonary thromboembolism; upper or lower extremity fracture in the past 3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 12-weeks in the Short Physical Performance Battery (SPPB) score | From baseline (T0) to 12-weeks (T2)
  Short Physical Performance Battery score measuring balance, lower extremity strength, and functional capacity in older adults. Minimum 0, maximum 12 (best)
Change from baseline to 6-weeks in the Short Physical Performance Battery (SPPB) score | From baseline (T0) to 6-weeks (T1)
  Short Physical Performance Battery score measuring balance, lower extremity strength, and functional capacity in older adults. Minimum 0, maximum 12 (best)
Change from 12-weeks to 24-weeks in the Short Physical Performance Battery (SPPB) score | From 12-weeks (T2) to 24-weeks (T3)
  Short Physical Performance Battery score measuring balance, lower extremity strength, and functional capacity in older adults. Minimum 0, maximum 12 (best)

SECONDARY OUTCOMES:
Change from baseline to 12-weeks in the Montreal Cognitive Assessment (MoCA) score | From baseline (T0) to 12-weeks (T2)
  Cognitive function (memory, language, attention, executive function, visuospatial and orientation). Minimum 0, maximum 30 (best)
Change from baseline to 6-weeks in the Montreal Cognitive Assessment (MoCA) score | From baseline (T0) to 6-weeks (T1)
  Cognitive function (memory, language, attention, executive function, visuospatial and orientation). Minimum 0, maximum 30 (best)
Change from 12 to 24-weeks in the Montreal Cognitive Assessment (MoCA) score | From 12-weeks (T2) to 24-weeks (T3)
  Cognitive function (memory, language, attention, executive function, visuospatial and orientation). Minimum 0, maximum 30 (best)
Change from baseline to 12-weeks in the Geriatric Depression Scale (GDS-15) | From baseline (T0) to 12-weeks (T2)
  Depressive symptoms measured with the Geriatric Depression Scale (GDS-15), minimum 0, maximum 15 (worse)
Change from baseline to 6-weeks in the Geriatric Depression Scale (GDS-15) | From baseline (T0) to 6-weeks (T1)
  Depressive symptoms measured with the Geriatric Depression Scale (GDS-15), minimum 0, maximum 15 (worse)
Change from 12-weeks to 24-weeks in the Geriatric Depression Scale (GDS-15) | From 12 weeks (T2) to 24-weeks (T3)
  Depressive symptoms measured with the Geriatric Depression Scale (GDS-15), minimum 0, maximum 15 (worse)
Change from baseline (T0) to 12-weeks (T2) in the Mini-Nutritional Assessment -Short Form (MNA-SF) | From baseline (T0) to 12-weeks (T2)
  Risk of malnutrition measured with the Mini-Nutritional Assessment -Short Form (MNA-SF), minimum 0, maximum 14 (best)
Change from baseline (T0) to 6-weeks (T1) in the Mini-Nutritional Assessment -Short Form (MNA-SF) | From baseline (T0) to 6-weeks (T1)
  Risk of malnutrition measured with the Mini-Nutritional Assessment -Short Form (MNA-SF), minimum 0, maximum 14 (best)
Change from 12-weeks (T2) to 24-weeks (T3) in the Mini-Nutritional Assessment -Short Form (MNA-SF) | From 12-weeks (T2) to 24-weeks (T3)
  Risk of malnutrition measured with the Mini-Nutritional Assessment -Short Form (MNA-SF), minimum 0, maximum 14 (best)
Change in the isometric handgrip strength from baseline (T0) to 12-weeks (T2) | From baseline (T0) to 12-weeks (T2)
  Best attempt of the isometric handgrip strength (kg) of the dominant hand evaluated by a hand-held dynamometer
Change in the isometric handgrip strength from baseline (T0) to 6-weeks (T1) | From baseline (T0) to 6-weeks (T1)
  Best attempt of the isometric handgrip strength (kg) of the dominant hand evaluated by a hand-held dynamometer
Change in the isometric handgrip strength from 12-weeks (T2) to 24-weeks (T3) | From 12-weeks (T2) to 24-weeks (T3)
  Best attempt of the isometric handgrip strength (kg) of the dominant hand evaluated by a hand-held dynamometer
Change in visual capacity from baseline (T0) to 12-weeks (T2) | From baseline (T0) to 12-weeks (T2)
  Distance and near vision assessed with WHO simple eye charts
Change in visual capacity from baseline (T0) to 6-weeks (T1) | From baseline (T0) to 6-weeks (T1)
  Distance and near vision assessed with WHO simple eye charts
Change in visual capacity from 12-weeks (T2) to 24-weeks (T3) | From 12-weeks (T2) to 24-weeks (T3)
  Distance and near vision assessed with WHO simple eye charts
Change in hearing capacity from baseline (T0) to 12-weeks (T2) | From baseline (T0) to 12-weeks (T2)
  HearWHO App consisting of an automated digit-in-noise test
Change in hearing capacity from baseline (T0) to 6-weeks (T1) | From baseline (T0) to 6-weeks (T1)
  HearWHO App consisting of an automated digit-in-noise test
Change in hearing capacity from 12-weeks (T2) to 24-weeks (T3) | From 12-weeks (T2) to 24-weeks (T3)
  HearWHO App consisting of an automated digit-in-noise test

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Jose Gimenez, PhD, Principal Investigator — European University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- See also: The Vivifrail multicomponent exercise program - Home page — http://vivifrail.com/